CLINICAL TRIAL: NCT00618670
Title: Home-based vs. Supervised Exercise for Claudicants
Brief Title: Home-based vs. Supervised Exercise for People With Claudication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Center for the Advancement of Science and Technology (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AG0095; R01AG024296 (NIH)
Record Dates: First submitted 2008-02-15; First posted 2008-02-20 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Intermittent Claudication
Keywords: aging; gait; musculoskeletal disorder therapy; peripheral blood vessel disorder; muscle function; muscle strength; quality of life
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Home-based program with progressive increases in exercise duration and intensity (i.e., cadence); walking duration will be longer for the home-based group because the intensity of walking will be lower than the graded treadmill walking performed by the supervised group
  Interventions: Behavioral: Walking Exercise
- 2 (Experimental): Supervised program consisting of graded treadmill walking, with progressive increments in exercise duration from 15 to 40 minutes, and progressive increments in exercise intensity from 50 to 70% of exercise capacity
  Interventions: Behavioral: Walking Exercise
- 3 (Active Comparator): Light resistance training without any walking exercise
  Interventions: Behavioral: Control--Resistance Training

INTERVENTIONS:
Behavioral: Walking Exercise — Three times per week for 3 months
  Arms: 1; 2
Behavioral: Control--Resistance Training — Three times per week for 3 months
  Arms: 3

SUMMARY:
The purpose of this study is to examine the effects of a home-based exercise rehabilitation program compared to a supervised exercise program on intermittent claudication (leg pain or discomfort) and ambulatory function.

DETAILED DESCRIPTION:
This study seeks to 1) compare the changes in ambulatory function, vascular function, and health-related quality of life in patients limited by intermittent claudication following a home-based exercise rehabilitation program, a supervised exercise program, and a light resistance training exercise program; and 2) determine whether changes in walking efficiency, calf muscle circulation, and calf muscle oxygen are the reasons by which both home-based and supervised exercise rehabilitation improve ambulatory function.

We hypothesize that a home-based exercise program utilizing new physical activity monitoring technology that can accurately quantify exercise adherence as well as the intensity, duration, and volume of exercise sessions will result in similar changes in ambulatory function, vascular function, and health-related quality of life compared to a standard, supervised exercise program. Further, both the home-based and supervised exercise rehabilitation programs will result in greater changes in ambulatory function, vascular function, and health-related quality of life than a light resistance training exercise program. Finally, we hypothesize that the changes in walking efficiency, calf muscle circulation, and calf muscle oxygen will each be predictive of improved ambulation following the home-based exercise program as well as the supervised exercise program.

The 3-month program will consist of walking 3 times per week, with progressive increases in duration and intensity. The two walking exercise programs will be matched on the estimated caloric expenditure during the training sessions. Patients in the control group will perform light resistance training without any walking exercise.

ELIGIBILITY:
Inclusion Criteria:

* Positive history of intermittent claudication assessed by the San Diego Claudication Questionnaire
* Exercise limited by intermittent claudication during a screening treadmill test using the Gardner protocol
* Ankle/brachial index (ABI) less than 0.90 at rest, which decreases to less than 0.73 immediately following the treadmill exercise test

Exclusion Criteria:

* Absence of PAD (peripheral artery disease)
* Asymptomatic PAD (Fontaine stage I)
* Rest pain due to PAD (Fontaine stage III)
* Tissue loss due to PAD (Fontaine stage IV)
* Medical conditions that are contraindicative for exercise according to the American College of Sports Medicine (e.g., acute myocardial infarction, unstable angina, etc.)
* Cognitive dysfunction (mini-mental state examination score less than 24)

Ages: 35 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in the walking distance to onset of leg pain, and the change in walking distance to maximal leg pain | 3 months

SECONDARY OUTCOMES:
Change in walking efficiency | 3 months
Change in calf muscle circulation and calf muscle oxygen | 3 months
Change in health-related quality of life | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Gardner, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- General Clinical Research Center, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Gardner AW, Poehlman ET. Exercise rehabilitation programs for the treatment of claudication pain. A meta-analysis. JAMA. 1995 Sep 27;274(12):975-80. PMID 7674529
- [Background] Gardner AW, Katzel LI, Sorkin JD, Bradham DD, Hochberg MC, Flinn WR, Goldberg AP. Exercise rehabilitation improves functional outcomes and peripheral circulation in patients with intermittent claudication: a randomized controlled trial. J Am Geriatr Soc. 2001 Jun;49(6):755-62. doi: 10.1046/j.1532-5415.2001.49152.x. PMID 11454114
- [Background] Gardner AW, Katzel LI, Sorkin JD, Goldberg AP. Effects of long-term exercise rehabilitation on claudication distances in patients with peripheral arterial disease: a randomized controlled trial. J Cardiopulm Rehabil. 2002 May-Jun;22(3):192-8. doi: 10.1097/00008483-200205000-00011. PMID 12042688
- [Background] Gardner AW, Killewich LA, Montgomery PS, Katzel LI. Response to exercise rehabilitation in smoking and nonsmoking patients with intermittent claudication. J Vasc Surg. 2004 Mar;39(3):531-8. doi: 10.1016/j.jvs.2003.08.037. PMID 14981444
- [Background] Gardner AW, Montgomery PS, Flinn WR, Katzel LI. The effect of exercise intensity on the response to exercise rehabilitation in patients with intermittent claudication. J Vasc Surg. 2005 Oct;42(4):702-9. doi: 10.1016/j.jvs.2005.05.049. PMID 16242558
- [Derived] Gardner AW, Montgomery PS, Wang M, Liang M. Effects of Long-Term Home Exercise in Participants With Peripheral Artery Disease. J Am Heart Assoc. 2023 Nov 7;12(21):e029755. doi: 10.1161/JAHA.122.029755. Epub 2023 Nov 6. PMID 37929770
- [Derived] Gardner AW, Parker DE, Montgomery PS. Changes in vascular and inflammatory biomarkers after exercise rehabilitation in patients with symptomatic peripheral artery disease. J Vasc Surg. 2019 Oct;70(4):1280-1290. doi: 10.1016/j.jvs.2018.12.056. Epub 2019 Mar 25. PMID 30922751
- [Derived] Gardner AW, Parker DE, Montgomery PS. Predictors of Improved Walking after a Supervised Walking Exercise Program in Men and Women with Peripheral Artery Disease. Int J Vasc Med. 2016;2016:2191350. doi: 10.1155/2016/2191350. Epub 2016 Dec 25. PMID 28116164
- [Derived] Gardner AW, Parker DE, Montgomery PS. Sex-specific predictors of improved walking with step-monitored, home-based exercise in peripheral artery disease. Vasc Med. 2015 Oct;20(5):424-31. doi: 10.1177/1358863X15596237. Epub 2015 Aug 3. PMID 26240075
- [Derived] Gardner AW, Parker DE, Montgomery PS, Blevins SM. Step-monitored home exercise improves ambulation, vascular function, and inflammation in symptomatic patients with peripheral artery disease: a randomized controlled trial. J Am Heart Assoc. 2014 Sep 18;3(5):e001107. doi: 10.1161/JAHA.114.001107. PMID 25237048
- [Derived] Gardner AW, Alaupovic P, Parker DE, Montgomery PS, Esponda OL, Casanegra AI. Influence of peripheral artery disease and statin therapy on apolipoprotein profiles. Int J Vasc Med. 2013;2013:548764. doi: 10.1155/2013/548764. Epub 2013 Sep 11. PMID 24102029
- [Derived] Gardner AW, Parker DE, Montgomery PS, Scott KJ, Blevins SM. Efficacy of quantified home-based exercise and supervised exercise in patients with intermittent claudication: a randomized controlled trial. Circulation. 2011 Feb 8;123(5):491-8. doi: 10.1161/CIRCULATIONAHA.110.963066. Epub 2011 Jan 24. PMID 21262997